CLINICAL TRIAL: NCT06787859
Title: Investigation of the Effect of "Curtain" Use on Self-Injection, Testing Fear and Pain in Patients With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hamdiye ARDA SÜRÜCÜ, Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICLE-ARDASURUCU-001
Record Dates: First submitted 2024-12-27; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus 2; Insulin Dependent Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, insulin, fear, pain,; curtain; Self-Injection
MeSH Terms: conditions — Diabetes Mellitus, Noninsulin-Dependent, 2; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Insulin Resistance; Pain

STUDY DESIGN:
Intervention Model Description: study group and control group
Who Masked: Participant
Masking Description: They do not know the experimental or control procedures that take place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental groups (Experimental): Nature-content "Curtain" will be shown before and during insulin injection administration
  Interventions: Other: Showing a nature view curtain to type 2 diabetic patients during insulin injection
- Nature-content "Curtain" Free (No Intervention): patients without of experimental Nature-content "Curtain"

INTERVENTIONS:
Other: Showing a nature view curtain to type 2 diabetic patients during insulin injection — a nature view curtain
  Arms: the experimental groups

SUMMARY:
Diabetes is a global problem for the world and negatively affects life (1). The most important reasons for ineffective diabetes and insulin treatment include fear of insulin side effects, fear of insulin injection, social embarrassment from administering insulin, fear of hypoglycemia and/or hyperglycemia (2). A large portion of diabetic individuals experience these fears, and some of these patients cope with these fears and integrate them into their daily lifestyles. However, some diabetic patients may be ineffective in coping with these fears (3). This situation creates negativities in the individual's success in treatment and compliance with treatment (3). Diverting attention is one of the non-pharmacological methods used in pain control. Diverting attention is one of the most preferred methods in reducing the pain experienced by patients during diagnosis and treatment procedures. It is a method that allows patients to control and reduce their symptoms by focusing their attention on a different point (4). In this study, the use of a distracting curtain during self-injection in individuals with Type 2 diabetes will be examined in order to examine the effect of pain and fear.

DETAILED DESCRIPTION:
Research Type:

It is designed as a randomized controlled, regular research.

Research Universe and Samples:

The research groups will be the living diabetes cells of Dicle University Hospitals. The research aims to create 100 healthy diabetes patients in Dicle University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least one year
* self-administering insulin injections
* self-administering a glucometer, insulin pen or insulin pump,

Exclusion Criteria:

* poor mental health
* Having gestational diabetes mellitus or Type 1 Diabetes

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale -VAS | Before insulin administration on day one Time Frame: After two insulin administration on the second day
  The VAS scale is used to assess subjectively perceived pain. The VAS scale is a 10 cm (100 mm) ruler with no pain at one end and "the most severe pain" at the other end. The individuals participating in the study were asked to mark the intensity of the pain they felt at that moment by explaining that the number "0" on the scale means "I do not feel any pain" and that the pain intensity increases as the numbers increase and that the number "10" means "I feel the most severe pain". In the evaluation, an increase in the score obtained from the scale indicates an increase in pain. It will be administered before and after each insulin injection. Each patient will be administered three times.

SECONDARY OUTCOMES:
Diabetes Fear of Self Injecting and Self-testing Questionnaire-D-FISQ | Before insulin administration on day one Time Frame: After two insulin administration on the second day
  The D-FISQ consists of two subscales: fear of self-injection (fear of self-injecting-FSI, 6 statements) and fear of self-testing (fear of self-testingFST, 9 statements). Each statement has a four-point Likert-type scale ranging from 0 to 3 (0= almost never, 1= sometimes, 2= often, 3= almost always). The evaluation of the questionnaire can be done by taking the average or raw score for the two sub-dimensions and the whole questionnaire. When taken as raw score, self-injection fear score ranges between 0-18, self-testing fear score ranges between 0-27, and total fear score ranges between 0-45. An increase in score indicates an increase in fear.
  It will be administered before and after each insulin injection. Each patient will be administered three times.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle Univertsity, Diyarbakır, South East, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No